CLINICAL TRIAL: NCT04414410
Title: Echocardiography in Critically-ill Patients With COVID-19 Pneumonia
Acronym: ECHO-COVID
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Prof Antoine Vieillard-Baron, Professor, Hospital Ambroise Paré Paris
Other Study IDs: RedCap19
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: COVID; Sars-CoV2
Keywords: critical care echocardiography; COVID; pneumonia; ICU
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Critical care echocardiography (CCE) has been widely used since the 10 last years. Covid outbreak leads that many patients with acute respiratory failure were admitted in the ICU. Many of these patients were ventilated and developed ARDS. Some of them developed deep vein thrombosis and pulmonary embolism. Nothing is already described about the cardiac function and the hemodynamics in these patients (how many RV failure, LV systolic dysfunction,...). The echo group of the cardiodynamix section of European society of intensive care medicien (ESICM) aims to promote CCE and evaluate its interest. The objective is to retrospectively enter in an international database all the echo studies done as usual care in these patients to evaluate (i) incidence of RV failure, (ii) incidence of LV systolic function, (iii) incidence of other patterns. Another objective will be to look for any association between some patterns and respiratory strategy, blood gas analysis, systemic hemodynamics. The echo studies were done and will be reported following one of the recent systematic review published by the same group (Huang S et al. AOIC 2020).

DETAILED DESCRIPTION:
Multicenter, international observational retrospective study. Patients admitted in the ICU between March 1th and april 26th for a pneumonia related to SARS COV 2 and who had at least one echocardiography during their stay will be included. Analysis will be retrospective in order to report the hemodynamic profile with left ventricular and right ventricular function. Will be also reported the respiratory settings, the central venous presure if available as well as usual parameters of macrocirculation. All data will be reported in RedCap by the University of sydney (https://redcap.sydney.edu.au/).

ELIGIBILITY:
Inclusion Criteria: patients admitted in the ICU for pneumonia related to SARS COV2 and who had at least 1 critical care echocardiography during the first 28 days.

-

Exclusion Criteria: Patients who did not have any critical care echocardiography during the first 28 days of the ICU stay.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: COVID 19 patients admitted in the ICU for respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Left ventricular systolic dysfunction | Up to 28 days
  LV systolic dysfunction is defined as an ejection fraction < 45%
Incidence of RV failure | up to 28 days
  RV failure is defined as RV/LV end-diastolic area > 0.8
Incidence of Vasoplegia | Up to 28 days
  Vasoplegia is defined as a normal or supranormal LV ejection fraction without echocarduiographic signs of hypovolemia.
Incidence of Hypovolemia | Up to 28 days
  Hypovolemia is defined as inspiratory collaspe of the superior vena cava in ventilated patients or virtual inferior vena cava in spontaneously breathing patients.

SECONDARY OUTCOMES:
Relation between plateau pressure and RV failure | Up to 28 days
  Plateau pressure and RV size
Relation between tidal volume and RV failure | Up to 28 days
  Tidal volume and RV size
Relation between PaO2 and RV failure | Up to 28 days
  PaO2, PaO2/FiO2, and RV size
Relation between PaCO2 and RV failure | Up to 28 days
  PaCO2 and RV size
Relation between PEEP and RV failure | Up to 28 days
  PEEP and RV size

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Vieillard-Baron, MD, PhD, Principal Investigator — Hospital Ambroise Paré Paris
Locations (1):
- University Hospital Ambroise Pare, Boulogne-Billancourt, Hauts De Seine, France

REFERENCES:
- [Derived] Huang S, Vieillard-Baron A, Evrard B, Prat G, Chew MS, Balik M, Clau-Terre F, De Backer D, Mekontso Dessap A, Orde S, Morelli A, Sanfilippo F, Charron C, Vignon P; ECHO-COVID study group. Echocardiography phenotypes of right ventricular involvement in COVID-19 ARDS patients and ICU mortality: post-hoc (exploratory) analysis of repeated data from the ECHO-COVID study. Intensive Care Med. 2023 Aug;49(8):946-956. doi: 10.1007/s00134-023-07147-z. Epub 2023 Jul 12. PMID 37436445